CLINICAL TRIAL: NCT05701488
Title: A Phase 1 Neoadjuvant Trial of Selective Internal Yttrium-90 Radioembolization (SIRT) With Tremelimumab and Durvalumab (MEDI4736) for Resectable Hepatocellular Carcinoma
Brief Title: SIRT With Tremelimumab and Durvalumab for Resectable HCC
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Jiping Wang, MD, PhD (Other)
Collaborators: AstraZeneca (Industry); Sirtex Medical (Industry)
Responsible Party: Sponsor-Investigator, Jiping Wang, MD, PhD, Principal Investigator, Dana-Farber Cancer Institute
Organization: Dana-Farber Cancer Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22-401
Record Dates: First submitted 2023-01-18; First posted 2023-01-27 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Resectable Hepatocellular Carcinoma; Hepatocellular Carcinoma; Hepatocellular Cancer
Keywords: Resectable Hepatocellular Carcinoma; Hepatocellular Carcinoma; Hepatocellular Cancer; Liver Cancer
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms | interventions — durvalumab; tremelimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Durvalumab + Tremelimumab (Arm A) (Experimental): -Participants will be randomized into the treatment group in a 1:1 ratio and will receive interventions as outlined:
  Neoadjuvant Treatment:
  * Cycle 1:
    * Day 1 of 28 Day Cycle: Pre-determined dose of Durvalumab and Tremelimumab
    * Day 28 of 28 Day cycle: Pre-determined dose of Durvalumab
  * Participants will undergo surgery on day 49 of Cycle 1. Surgery will be performed per institutional standard of care.
  Adjuvant Treatment:
  --Cycles 1 (28 days postoperatively) - 13:
  ---Day 1 of 28 Day Cycle: Pre-determined dose of Durvalumab
  Interventions: Drug: Durvalumab; Drug: Tremelimumab
- Durvalumab + Tremelimumab + SIRT (Arm B) (Experimental): -Participants will be randomized into the treatment group in a 1:1 ratio and will receive interventions as outlined:
  Neoadjuvant Treatment:
  * Cycle 1:
    * Day 3 of 28 Day Cycle: Pre-determined dose of Durvalumab and Tremelimumab
    * Day 31 of 28 Day Cycle: Pre-determined dose of Durvalumab
    * Day 1 of 28 Day Cycle: Yttrium-90
  * Participants will undergo surgery on Day 52 of Cycle 1. Surgery will be performed per institutional standard of care.
  Adjuvant Treatment:
  --Cycles 1 (28 days postoperatively) - 13:
  ---Day 1 of 28 Day Cycle: Pre-determined dose of Durvalumab
  Interventions: Drug: Durvalumab; Drug: Tremelimumab; Device: SIRT

INTERVENTIONS:
Drug: Durvalumab — Intravenous infusion
  Other Names: Imjudo; MEDI4736
Drug: Tremelimumab — Intravenous infusion
  Other Names: Imfinzi
Device: SIRT — SIR (Selective Internal Radiation) Sphere resin microspheres, radioactive particles delivered via injection into an artery.
  Other Names: Selective Internal Yttrium-90 Radioembolization
  Arms: Durvalumab + Tremelimumab + SIRT (Arm B)

SUMMARY:
The goal of this research study is to evaluate the safety and tolerability of tremelimumab and durvalumab with or without Selective Internal Yttrium-90 Radioembolization (SIRT) in participants with resectable hepatocellular carcinoma (HCC) who will undergo liver surgery.

The names of the interventions involved in this study are:

* Durvalumab (a type of immunotherapy)
* Tremelimumab (a type of immunotherapy)
* Selective Internal Yttrium-90 Radioembolization (SIRT) (a type of radiation microsphere bead)

DETAILED DESCRIPTION:
This is a Phase 1, open-label, randomized research study to evaluate the safety and tolerability of tremelimumab and durvalumab with or without Selective Internal Yttrium-90 Radioembolization (SIRT) in participants with resectable hepatocellular carcinoma (HCC) who will undergo liver surgery.

Participants will be randomized into one of two treatment groups: Durvalumab + Tremelimumab versus Durvalumab + Tremelimumab + SIRT. Randomization means that a participant is put into a group by chance. Radioembolization is a combination of radiation therapy and a procedure called embolization to treat cancer. SIRT blocks tumor blood supply by injecting radioactive particles into the hepatic artery and delivers internal radiotherapy on the tumor.

The U.S. Food and Drug Administration (FDA) has not approved Durvalumab as treatment for HCC but it has been approved for other uses.

The U.S. FDA has not approved tremelimumab as a treatment option for HCC.

The research study procedures include screening for eligibility, study treatment including evaluations, radiology scans of the liver, blood tests, electrocardiograms, and follow up visits.

Participation in this study is expected to last about 18 months with long-term follow up for a maximum of 3 years.

It is expected that about 20 people will take part in this research study.

AstraZeneca, a pharmaceutical company, is supplying the study drugs, tremelimumab and durvalumab. Sirtex Medical Inc., a medical device company, is supplying the Yttrium-90 resin Microsphere beads.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed HCC (documentation of original biopsy for diagnosis is acceptable if tumor tissue is unavailable) or clinical diagnosis by American Association for the Study of Liver Diseases (AASLD) criteria in cirrhotic subjects (presence of arterial hypervascularity with venous washout). For subjects without cirrhosis, histological confirmation is mandatory.
* Participants must have resectable disease. Those patients must have preserved liver function (Child A) and with either AJCC stage IA, IB, II, and IIIA or BCLC stage 0 or stage A disease. The determination of resectability will ultimately lie in the clinical judgment of the treating investigator and surgical oncologist involved in the care of the patient.
* Participants must be treatment naïve for HCC.
* Age ≥18 years. Because no dosing or adverse event data are currently available on the use of tremelimumab, durvalumab, and SIRT in participants <18 years of age, children are excluded from this study.
* Measurable disease per RECIST 1.1 criteria.
* ECOG performance status ≤ 1 (see Appendix A).
* Body weight >30 kg.
* Participants must have adequate organ and marrow function as defined below:

  * Hemoglobin ≥ 9.0 g/dL
  * Absolute Neutrophil Count (ANC) ≥ 1,000 /mcL
  * Platelets ≥ 80,000 /mcL
  * Total Bilirubin ≤ 2.0 mg/dL
  * AST (SGOT) and ALT (SGPT) ≤ 2.5 × institutional upper limit of normal (ULN)
  * Measured Creatinine Clearance > 40 mL/min by 24-hour urine collection, or
  * Calculated Creatinine Clearance (CL) > 40 mL/min by the Cockcroft-Gault Formula (Cockcroft Gault 1976):

    * Males: Creatinine CL (mL/min) = (weight (kg) × (140 - Age)) / (72 × serum creatinine (mg/dL))
    * Females: Creatinine CL (mL/min) = (weight (kg) × (140 - Age) / (72 × serum creatinine (mg/dL))) × 0.85
* Women of childbearing potential (WOCBP, refer to Section 5.4) must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropin [HCG]) obtained during the trial screening period.
* Men and WOCBP must agree to follow the protocol instructions for acceptable method(s) of contraception for the duration of trial treatment and for a total of 5 months post-treatment completion. Refer to Section 5.4.
* Participants with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen as assessed by the treating investigator are eligible for this trial.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Participants who have received any prior treatment for HCC.
* Patients who have had a major surgical procedure, open biopsy, or significant traumatic injury with poorly healed wound within 6 weeks prior to first dose of study drug.
* History of allogenic organ transplantation.
* Participants who are receiving any other investigational agents.
* Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc.]). The following are exceptions to this criterion:

  * Patients with vitiligo or alopecia
  * Patients with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement
  * Any chronic skin condition that does not require systemic therapy
  * Patients with celiac disease controlled by diet alone
  * Patients without active disease in the last 5 years may be included but only after consultation with the sponsor-investigator
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to durvalumab or tremelimumab.
* Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection (including tuberculosis), uncontrolled hypertension (defined as blood pressure of > 140/90 mmHg during the screening period despite medical management), interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs, or compromise the ability of the patient to give written informed consent.
* Patients who have a primary brain tumor (excluding meningiomas and other benign lesions), any brain metastases, leptomeningeal disease, seizure disorders not controlled with standard medical therapy, or history of a stroke within the year prior to the first dose of study drug.
* History of active primary immunodeficiency.
* Known active infection of human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS)

  --Patients positive for HIV are allowed on study, but HIV-positive patients must have:
  * A stable regimen of highly active anti-retroviral therapy (HAART)
  * No requirement for concurrent antibiotics or antifungal agents for the prevention of opportunistic infections
  * A CD4 count above 250 cells/mcL and an undetectable HIV viral load or standard PCR-based tests
* Known active hepatitis B infection (known positive HBV surface antigen (HBsAg) result). Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible.
* Known active hepatitis C infection. Participants positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
* Current or prior use of immunosuppressive medication within 14 days before the first dose of study agent. The following are exceptions to this criterion:

  * Intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra-articular injection)
  * Systemic corticosteroids at physiologic doses that do not exceed 10 mg/day of prednisone or its equivalent
  * Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication)
* Receipt of live attenuated vaccine within 30 days prior to the first dose of study drug. Note: Patients, if enrolled, should not receive live vaccine whilst receiving study drug and for at least 30 days after the last dose of study agent.
* History of serious systemic disease, including myocardial infarction or unstable angina within the 12 months prior to the first dose of study drug, history of hypertensive crisis or hypertensive encephalopathy, New York Heart Association (NYHA) grade II or greater congestive heart failure, unstable symptomatic arrhythmia requiring medication (patients with chronic atrial arrhythmia, i.e., atrial fibrillation or paroxysmal supraventricular tachycardia are eligible), significant vascular disease or symptomatic peripheral vascular disease.
* Participants who have a known clinical history of coagulopathy, bleeding diathesis, or thrombosis within the 12 months prior to the first dose of study drug.
* Participants who have a serious, non-healing wound, ulcer, bone fracture or with history of pneumonitis or interstitial lung disease.
* Participants who are pregnant or breastfeeding. A negative serum or urine pregnancy test obtained during the screening period is required for trial enrollment.
* Participants requiring total parenteral nutrition with lipids.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-04-21 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events | up to 18 months
  Defined as All grade 3-5 adverse events (AE) with treatment attribution of possibly, probably or definite based on CTCAEv5 as reported on case report forms were counted. Rate is the proportion of treated participants experiencing at least one treatment-related grade 3-5 AE of any type during the time of observation.

SECONDARY OUTCOMES:
Best Radiologic Response | up to 15 months
  Defined as best radiologic response on treatment and evaluated per RECIST 1.1 criteria.
Best Pathological Response | up to 65 days
  Defined as the best pathological response based on evaluation of the surgical sample defined per protocol for gross and microscopic evaluation.
Median Overall Survival (OS) | up to 3 years
  Calculated via the Kaplan-Meier method and defined as the time from study entry to death or censored at date last known alive.
Median Progression-Free Survival (PFS) | up to 3 years
  Calculated via the Kaplan-Meier method and defined as the duration between randomization and documented disease progression or death, or is censored at time of last disease assessment.
CD8+/CD4+T Cells Level | up to 3 years
  Comparison between pre-treatment and post-treatment via paired t-test and Wilcoxon signed rank test and Fisher's exact test.
Dendritic Cells Level | up to 3 years
  Comparison between pre-treatment and post-treatment via paired t-test and Wilcoxon signed rank test and Fisher's exact test.
Cytokines Level | up to 3 years
  Comparison between pre-treatment and post-treatment via paired t-test and Wilcoxon signed rank test and Fisher's exact test. IL-1b, IL-2, IL-6, TNFa, IFNg, CCL2, IL-8, IL-18, CXCL9, CXCL10 will be measured by cytokine bead array and reported as picrograms per mL (pg/mL).
Number of Participants with Surgical Complications | up to 30 days
  Surgical complications will be defined by postoperative occurrences and defined according National Surgical Quality Improvement Program (NSQIP) criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Jiping Wang, MD, PhD, Principal Investigator — Dana-Farber Cancer Institute
Locations (3):
- United States (3):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: BWH - Contact the Partners Innovations team at http://www.partners.org/innovation